CLINICAL TRIAL: NCT01068899
Title: Energy Expenditure
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Aline Andres, Ph.D., University of Arkansas for Medical Sciences
Other Study IDs: 111597
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: healthy adults; healthy children

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children: healthy children
- Adult: healthy adults

SUMMARY:
The purpose of this study is to standardize methods in measuring a person's energy expenditure. These methods may be used in a larger study in the future.

ELIGIBILITY:
Inclusion Criteria:

* adults must be 18 years of age or older
* children must be between 6 and 88 pounds

Exclusion Criteria:

* pulmonary or respiratory disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy women and children who do not have any respiratory or pulmonary disorders
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States